CLINICAL TRIAL: NCT02306278
Title: The Effects of Gabapentin Premedication on Postoperative Pain,Nausea,Vomiting and Sedation in Patients Undergoing Neurosurgery
Brief Title: The Effects of Gabapentin Premedication on Neurosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Wei Zhang, attending doctor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ky2013-008-01
Record Dates: First submitted 2014-04-16; First posted 2014-12-03 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Cerebral Tumor
Keywords: gabapentin; postoperative pain; vomiting; nausea
MeSH Terms: conditions — Pain, Postoperative; Vomiting; Nausea | interventions — Gabapentin; Vitamins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin capsules (Placebo Comparator): vitamin capsules orally at the night before operation and 2 hours before surgery,respectively
  Interventions: Drug: vitamin capsules
- gabapentin (Experimental): gabapentin 600mg orally at the night before operation and 2 hours before surgery,respectively
  Interventions: Drug: gabapentin

INTERVENTIONS:
Drug: gabapentin — gabapentin capsules 0.3g
  Arms: gabapentin
Drug: vitamin capsules — vitamin B
  Arms: vitamin capsules

SUMMARY:
The study is to observe the effects of gabapentin premedication on postoperative pain,vomiting and nausea in patients undergoing neurosurgery. 100 neurosurgical patients are randomized into groups gabapentin(GG) or placebo(GP). Patients are given gabapentin or placebo orally the night before operation day and 2hours before surgery,respectively.The investigators hypothesized that lower incidence of postoperative pain,vomiting and nausea be observed in GG than GP.

DETAILED DESCRIPTION:
This is a random, double-blind study. In GG, patients are given gabapentin 600mg orally at the night and 2hours before surgery, respectively. In PG, vitamine pills are given instead.Total intravenous anesthesia is applied for all patients. 1hour, 2hours,1day, 2days, 3months and 6months after surgery, patients are evaluated for pain (VAS) and incidence of PONV. In addition,Glasgow Score, Ramsay Score and other gabapentin-related effects, such as somnolence,dizzy or dry mouth are also observed.The incidence of persistent pain and neuropathic pain was assessed at the 3-mo and 6-mo postoperative evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old, ASA physical status I or II, BMI<30
* Scheduled for elective craniotomy
* Cooperative and given informed consent in person

Exclusion Criteria:

* History of mental or psychiatric disorders
* Pregnant or lactating female
* History of systemic malignant tumor or diabetes
* Previously treated with this protocol or participated in another experimental study within previous 30 days
* Suspected history of allergic reaction or intolerance to gabapentin or other anesthetic agents in this study
* History of alcohol abuse and/or drug abuse within previous one year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2014-12-14 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Premedication gabapentin can decrease pain in early postoperative period | 24 hour after extubation
  postoperative pain scores(Visual Analogue Scale)

SECONDARY OUTCOMES:
Premedication gabapentin can limit the development of persistent pain and neuropathic pain. | 3-mos and 6-mos after surgery
  postoperative pain scores(Visual Analogue Scale) and the Leeds assessment of neuropathic symptoms and signs (LANSS) Pain Scale
Preoperative gabapentin can lead to a decrease incidence of PONV | 1 hour,2 hours,1day,2 days after surgery
  Incidence of PONV

OTHER OUTCOMES:
The gabapentin-related effects on neurosurgical patients | 1 hour,2 hours,1day,2 days after surgery
  Glasgow Score, Ramsay Score , somnolence,dizzy or dry mouth

CONTACTS AND LOCATIONS:
Overall Officials: Ru Quan Han, chief, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Department of Anesthesiology,Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China